CLINICAL TRIAL: NCT00515736
Title: Influence Of Early Antioxidant Supplements On Clinical Evolution And Organ Function In Critically Ill Cardiac Surgery, Major Trauma And Subarachnoid Hemorrhage Patients
Brief Title: Impact Of Antioxidant Micronutrients On Intensive Care Unit (ICU) Outcome
Acronym: Etude-AOX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: enrollment was completed
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Prof Mette M Berger, MD, PhD, Dept of Adult Intensive Care, CHUV
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CE-102-02
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2008-04

CONDITIONS: Critically Ill Patients; Cardiac Surgery; Trauma; Subarachnoid Hemorrhage
Keywords: selenium; oxidative stress; glutathione peroxidase; critically ill; outcome; supplementation
MeSH Terms: conditions — Wounds and Injuries; Subarachnoid Hemorrhage; Critical Illness | interventions — Selenium; Zinc; Ascorbic Acid; Thiamine; Vitamin E; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AOX group (Experimental): Treatment group - double dose (loading) for 48 hours then single dose (Se 270 mcg, Zn 30 mg, vit C 1.2 g, B1 100 mg, vit E 300 mg enteral)
  Interventions: Drug: Selenium (Se), Zinc (Zn), Vitamin C, Vitamin B1, Vitamin E
- 0 (Placebo Comparator): Group receiving vehicle solution for 5 days (double dose for 48 hours)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Selenium (Se), Zinc (Zn), Vitamin C, Vitamin B1, Vitamin E — Se 270mcg, Zn 30mg, C 1.1g, B1 100mg, E 300mg
  Other Names: Selenium - Laboratoire Aguettant; Zinc - Laboratoire Aguettant, the others generic
  Arms: AOX group
Drug: Placebo — vehicle
  Other Names: vehicle - NaCl 0.9% solution
  Arms: 0

SUMMARY:
Critically ill patients are generally exposed to an increased oxidative stress, which is proportional to the severity of their condition. Endogenous antioxidant (AOX) defenses are depleted particularly in those patients with intense inflammatory response. The hypothesis tested is that early I:V: administration of a combination of AOX micronutrient supplements (Se, Zn, Vit C, Vit E, Vit B1) would improve clinical outcome in selected critically ill patients, by reinforcing the endogenous AOX defenses and reducing organ failure.

DETAILED DESCRIPTION:
Prospective randomized, double-blind, placebo-controlled, single-center trial. Patients admitted to ICU after complicated cardiac surgery, major trauma with or without brain injury, subarachnoid hemorrhage, and predicted by the clinicians to require >48 hours of ICU treatment.

Supplements: provided IV for 5 days

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted for above diagnosis assessed on admission by the medical team likely to require more than 48 hours of ICU

Exclusion Criteria:

* absence of consent, participation in another study, liver cirrhosis or major burns and life expectancy < 24 hours or a lack of commitment to full aggressive care (anticipated withholding or withdrawing treatments in the 48 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Organ function (SOFA) with special additional attention to renal function | 3 months

SECONDARY OUTCOMES:
Pneumonia, Length of mechanical ventilation-ICU stay-hospital stay, Mortality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Berger, MD PhD, Principal Investigator — Dpt of Adult Intensive Care, CHUV
Locations (1):
- Dpt of Adult Intensive Care - CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Result] Berger MM, Soguel L, Shenkin A, Revelly JP, Pinget C, Baines M, Chiolero RL. Influence of early antioxidant supplements on clinical evolution and organ function in critically ill cardiac surgery, major trauma, and subarachnoid hemorrhage patients. Crit Care. 2008;12(4):R101. doi: 10.1186/cc6981. Epub 2008 Aug 7. PMID 18687132